CLINICAL TRIAL: NCT06385938
Title: Ultrasound Imaging and Quantitative Vibro-acoustic Assessment of Rickets in Children
Brief Title: Ultrasound Imaging and Quantitative Vibro-Acoustic Assessment of Rickets Under the Age of Ten
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas Thacher, Principal Investigator, Mayo Clinic
Other Study IDs: 23-012048
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Rickets
MeSH Terms: conditions — Rickets | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Active Rickets Group: Children under 10 years of age with a diagnosis of active rickets on radiographs of the wrists and knees will undergo ultrasound imaging and quantitative vibro-acoustic assessment.
  Interventions: Diagnostic Test: Ultrasound with quantitative vibro-acoustic assessment
- Healthy Children Control Group: Healthy children under 10 years of age not diagnosed with rickets, but match the age, gender, and weight of the children with rickets, will undergo ultrasound imaging and quantitative vibro-acoustic assessment.
  Interventions: Diagnostic Test: Ultrasound with quantitative vibro-acoustic assessment

INTERVENTIONS:
Diagnostic Test: Ultrasound with quantitative vibro-acoustic assessment — Imaging with non-invasive bone assessment based on wide range of frequencies and free from soft tissue artifact of the wrists and the knees

SUMMARY:
The goal of this study is to find out if the use of ultrasound pictures of bones can spot changes in the growth areas of children with rickets, a condition that affects how bones harden. Researchers want to see if these ultrasound pictures can help tell the difference between children who have rickets and those who don't.

DETAILED DESCRIPTION:
Aims, purpose, or objectives:

1. To determine if ultrasound imaging of bone can identify the changes of impaired mineralization of the growth plates at the wrists and the knees, similar to those visible on plain radiographs.
2. To determine if quantitative vibro-acoustic measurements of the bone in subjects with rickets significantly differs from control subjects, matched for age, sex, and BMI.
3. To determine the relationship of ultrasound images and quantitative vibro-acoustic assessment with rickets severity score (RSS), based on radiographs of the wrists and knees.
4. To determine if longitudinal changes in ultrasound images and quantitative vibro-acoustic assessment with treatment of rickets are related to changes in the rickets severity score.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Prepubertal children less than 10 years of age with active nutritional or genetic rickets at enrollment (RSS>1.5 based on radiographs of the wrists and knees performed within 3 months prior to enrollment). Cases will be recruited from the Pediatric Endocrinology Bone Clinic or from the Mayo Clinic outpatient or inpatient services in Rochester, MN. Cases who return for follow-up and demonstrate improvement in RSS≥1.0 will be eligible for a single repeat ultrasound evaluation.
* Controls: Healthy children empaneled in Mayo Clinic primary care (Family Medicine or Community Pediatrics) matched for age (±3 months), sex, and BMI (±0.5 kg/m2)

Exclusion Criteria:

* Known fracture at imaging site
* Rickets of prematurity

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prepubertal children <10 years of age at enrollment with active nutritional or genetic rickets recruited from the Mayo Clinic Pediatric Endocrinology Bone Clinic or from the Mayo Clinic outpatient or inpatient services in Rochester, MN (cases). Healthy matched control children will be recruited from children empaneled in Mayo Clinic primary care (Family Medicine or Community Pediatrics).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Relationship of quantitative vibro-acoustic ultrasound and rickets severity score | Baseline
  Quantitative vibro-acoustic data will be compared with the radiographic rickets severity score to assess if ultrasound measures are reliably related to the radiographic findings.

SECONDARY OUTCOMES:
Relationship of ultrasound images with radiographic evidence of rickets | Baseline
  Determine if ultrasound imaging of bone can identify the changes of impaired mineralization of the growth plates at the wrists and the knees, similar to those visible on plain radiographs
Case-control comparison of quantitative vibro-acoustic ultrasound measurements between children with rickets and control subjects | Baseline
  2. To determine if quantitative vibro-acoustic measurements of the bone in subjects with rickets significantly differs from control subjects, matched for age, sex, and BMI.
Longitudinal changes in vibro-acoustic ultrasound measurements with treatment of rickets | Baseline
  To determine if longitudinal changes in ultrasound images and quantitative vibro-acoustic assessment with treatment of rickets are related to changes in the rickets severity score

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Thacher, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials